CLINICAL TRIAL: NCT02059629
Title: Eluna Family / Sentus BP Master Study
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: CR014
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Bradycardia; Heart Failure
Keywords: Heart failure; Eluna pacemaker family; Sentus OTW BP L left ventricular lead; Bradycardia; SADE-free rate
MeSH Terms: conditions — Bradycardia; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Eluna pacemaker family: Patients with standard indication for pacemaker therapy or Cardiac Resynchronization Therapy (CRT), who will be implanted with a pacemaker or CRT device of the Eluna pacemaker family. Single-, Dual- and Tripple-chamber pacemakers are applicable.
  Interventions: Device: Eluna pacemaker family
- Group B: Sentus BP lead: Heart failure patients with indication for Cardiac Resynchronization Therapy (CRT) therapy, who will be implanted with the left ventricular Sentus BP lead. Patients can receive either CRT pacemaker or CRT-D (CRT with defibrillator function).
  Interventions: Device: Sentus BP lead

INTERVENTIONS:
Device: Eluna pacemaker family — New pacemaker generation with new functions, like wandless RF telemetry "SafeSync"
  Other Names: Eluna SR-T/DR-T/HF-T; Etrinsa SR-T/DR-T/HF-T; Epyra SR-T/DR-T/HF-T
  Groups: Group A: Eluna pacemaker family
Device: Sentus BP lead — over-the-wire (OTW), bipolar (BP), L-shaped (L), 4.8 French left ventricular lead
  Other Names: Sentus OTW BP L
  Groups: Group B: Sentus BP lead

SUMMARY:
The Eluna Family / Sentus BP Master Study is designed to confirm the safety of the new Eluna pacemaker family and the Sentus BP (bipolar) left ventricular lead.

Furthermore the new wandless RF telemetry function "SafeSync" and the handling of the Sentus lead during implantation will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing to participate in the study and provided written informed consent
* Patient meets standard indication for pacemaker or CRT-P or CRT-D therapy
* Patient accepts Home Monitoring® concept
* Patient has legal capacity and ability to consent

Exclusion Criteria:

* Patient with any contraindication to pacemaker and CRT-P and CRT-D therapy
* Patient under the age of 18
* Pregnant or breast-feeding women
* Cardiac surgery planned within the next 6 months
* Life expectancy less than 12 months
* Participation in another cardiac clinical investigation with active treatment arm
* Group B only: Currently implanted with an endocardial or epicardial LV lead or had prior attempt to place a LV lead (for CRT implants only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from available pacemaker or CRT patients directly by the treating physician at the investigational site
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Eluna pacemaker family: Serious Adverse Device Effect (SADE) - free rate | 6 months
  The safety of the Eluna pacemaker family will be evaluated by asking the investigator to record any adverse event. While all adverse events have to be recorded throughout the study, only the number of SADEs possibly or securely related to the pacemaker will be the basis for endpoint calculation of the SADE-free rate.
Sentus BP lead: Serious Adverse Device Effect (SADE) - free rate | 3 months
  The safety of the Sentus BP left ventricular lead will be evaluated by asking the investigator to record any adverse event. While all adverse events have to be recorded throughout the study, only the number of SADEs possibly or securely related to the Sentus BP lead will be the basis for endpoint calculation of the SADE free rate.

OTHER OUTCOMES:
Collection of data of interest: Handling assessment of Sentus lead during implantation | 3 months
Collection of further data of interest: Evaluation of wandless RF telemetry function "SafeSync" in the Eluna pacemaker family | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Georges Mairesse, Dr. med, Principal Investigator — Cliniques du Sud Luxembourg
Locations (17):
- Allgemeines Krankenhaus Linz, Linz, Austria
- Belgium (2):
  - Cliniques du Sud Luxembourg, Arlon
  - ZOL Genk, Genk
- Denmark (3):
  - Aalborg Sygehus, Aalborg
  - Gentofte Hospital, Hellerup
  - Odense University Hospital, Odense
- Germany (10):
  - Charité Universitätsmedizin Berlin, CBF: Campus Benjamin Franklin, Berlin
  - Charité - Universitätsmedizin Berlin, CVK: Campus Virchow-Klinikum, Berlin
  - Klinikum Lippe, Detmold
  - Universitätsklinikum Erlangen, Medizinische Klinik 2, Erlangen
  - Universitätsklinikum Essen, Westdeutsches Herzzentrum Essen, Essen
  - Elisabeth Krankenhaus Essen, Essen
  - Universitäts-Herzzentrum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Greifswald, Greifswald
  - St. Marien-Hospital Lünen, Lünen
  - Marienhaus GmbH St. Elisabeth Krankenhaus Saarlouis, Saarlouis
- Queen Mary Hospital, Hong Kong, Hong Kong